CLINICAL TRIAL: NCT02584777
Title: A Phase II, Prospective, Non-Controlled, Open-Label, Efficacy, Safety, Pharmacokinetic, and Pharmacodynamic Study of Pacritinib in Asian Subjects With Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis or Post- Essential Thrombocythemia Myelofibrosis
Brief Title: A Phase II Non-Controlled, Open-Label, Efficacy, Safety, Pharmacokinetic, and Pharmacodynamic Study of Pacritinib in Myelofibrosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 381401
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Primary Myelofibrosis
Keywords: Post-essential thrombocythemia myelofibrosis; Post-Polycythemia Vera Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pacritinib (Experimental): Oral administration
  Interventions: Biological: Pacritinib

INTERVENTIONS:
Biological: Pacritinib — QD (Once a day)

SUMMARY:
To evaluate the efficacy, safety, pharmacokinetics (PK) and pharmacodynamics (PD) of pacritinib in Asian subjects with myelofibrosis (MF), which includes primary MF (PMF), post-polycythemia vera MF (PPV-MF) or post-essential thrombocythemia MF (PET-MF).

ELIGIBILITY:
Inclusion Criteria:

1. Intermediate-1, intermediate-2, or high-risk PMF, PPV-MF or PET-MF as based on The Dynamic International Prognostic Scoring System (DIPSS) criteria
2. Palpable splenomegaly ≥5 cm below the LCM in midclavicular line by physical examination
3. TSS ≥13 on the MPN-SAF TSS 2.0, not including the inactivity question, based on a single assessment during screening visit
4. Age ≥18 years old at the time of screening (or minimum age of legal consent consistent with local regulations, if minimum is >18 years of age)
5. ECOG performance status 0 to 3
6. Peripheral blast count <10%
7. Absolute neutrophil count >500/μL
8. Participants who are platelet or RBC transfusion dependent are eligible
9. Adequate liver and renal function, defined by liver transaminases (AST/serum glutamic oxaloacetic transaminase [SOOT] and alanine aminotransferase [ALT]/serum glutamic pyruvic transaminase [SGPT]) ≤3 × upper limit of normal ([ULN], AST/ALT ≤5 × ULN if transaminase elevation is related to MF), direct bilirubin ≤4 × ULN, and creatinine ≤2.5 mg/dL
10. At least 6 months from prior splenic irradiation
11. At least 12 months from prior 32P therapy
12. At least 1 week since prior treatment (most recent dose) with a potent CYP3A4 inhibitor or inducer
13. At least 4 weeks since any experimental treatment for PMF, PPV-MF, or PET-MF
14. At least 2 weeks since any treatment for PMF, PPV-MF, or PET-MF
15. If fertile, both males and females must agree to use effective birth control.
16. Able to understand and willing to complete symptom assessments using a patient-reported outcomes instrument and comply with treatment and study procedures of the protocol
17. Able to understand and willing to sign the informed consent form (ICF)
18. Participant is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

1. Any GI or metabolic condition that could interfere with absorption of oral medication
2. Life expectancy <6 months
3. Prior treatment with a JAK2 inhibitor
4. Completed ASCT, or are eligible for and willing to complete ASCT
5. History of splenectomy or planning to undergo splenectomy
6. Uncontrolled intercurrent illness, including but not limited to ongoing active infection, or psychiatric illness, or social situation that, in the judgment of the treating physician, would limit compliance with study requirements
7. Other malignancy within the last 3 years, other than curatively treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, organ confined, or treated non-metastatic prostate cancer with negative prostate specific antigen, in situ breast carcinoma after complete surgical resection, or superficial transitional cell bladder carcinoma
8. Inflammatory or chronic functional bowel disorder, such as Crohn's disease, inflammatory bowel disease, chronic diarrhea, or constipation
9. Clinically symptomatic and uncontrolled cardiovascular disease
10. History of any of the following within 6 months prior to first dose of pacritinib: myocardial infarction, severe/unstable angina, or symptomatic congestive heart failure
11. New York Heart Association Class II, III, or IV congestive heart failure
12. Participants with NCI CTCAE (version 4.03) Grade 2 cardiac arrhythmias may be considered for inclusion, with the approval of the medical monitor, if the arrhythmias are stable, asymptomatic and unlikely to affect participant safety. Participants will be excluded if they have ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥3, QTc prolongation >450 ms, or other conditions that increase the risk for QT interval prolongation (eg, heart failure, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], or family history of long QT interval syndrome)
13. Erythropoietic agent within 28 days prior to first dose of pacritinib
14. Thrombopoietic agent within 14 days prior to first dose of pacritinib
15. Known seropositivity for human immunodeficiency virus or syphilis, or known active hepatitis A, B or C virus infection
16. Participant has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
17. Participant is a family member or employee of the investigator
18. If female, participant is pregnant or breastfeeding at the time of enrollment. Even if breastfeeding can be discontinued, the participant should not be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving a ≥35% reduction in spleen volume | Baseline to Week 24
  Measured by MRI or CT scan

SECONDARY OUTCOMES:
Proportion of participants with ≥50% reduction in total symptom score (TSS) | Baseline to Week 24
  Measured by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) TSS 2.0
Proportion of participants with baseline platelet count <100,000/μL achieving ≥35% reduction in spleen volume | Baseline to Week 24
  Measured by MRI or CT scan
Proportion of participants with baseline platelet count <100,000/μL achieving ≥50% reduction in total symptom score (TSS) | Baseline to Week 24
Proportion of participants with baseline platelet count <50,000/μL achieving ≥35% reduction in spleen volume | Baseline to Week 24
  Measured by MRI or CT scan
Proportion of participants with baseline platelet count <50,000/μL achieving ≥50% reduction in total symptom score (TSS) | Baseline to Week 24
Clinically significant adverse events (AEs) | Throughout the study period of approximately 5 years
Clinically significant changes in laboratory results | Throughout the study period of approximately 5 years
Clinically significant changes in vital signs | Throughout the study period of approximately 5 years
Clinically significant changes in electrocardiograms (ECGs) | Throughout the study period of approximately 5 years
Pacritinib pharmacokinetic (PK) parameter: maximum observed concentration (Cmax) | Baseline; weeks 3, 12 & 24
Pacritinib pharmacokinetic (PK) parameter: Time of maximum observed concentration (Tmax) | Baseline; weeks 3, 12 & 24
Pacritinib pharmacokinetic (PK) parameter: minimum observed concentration (Cmin) | Baseline; weeks 3, 12 & 24
Pacritinib pharmacokinetic (PK) parameter: area under the concentration curve (AUC) | Baseline; weeks 3, 12 & 24
Pacritinib pharmacokinetic (PK) parameter: apparent volume of distribution (V/F) | Baseline; weeks 3, 12 & 24
Pharmacodynamic parameter: Maximum observed effect (Emax) | Baseline; weeks 3, 12 & 24
Pharmacodynamic parameter: time of maximum observed effect (tEmax) | Baseline; weeks 3, 12 & 24
Pharmacodynamic parameter: area under the effect curve (AUEC) | Baseline; weeks 3, 12 & 24

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda